CLINICAL TRIAL: NCT00691782
Title: The Impact of African American Women's Hair Care Practices and Hair Attitudes on Exercise Habits
Status: Completed | Type: Observational
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Other Study IDs: IRB00003923
Record Dates: First submitted 2008-06-02; First posted 2008-06-05 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Hair and Scalp Health
Keywords: African American females between the ages of 21 and 60

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: African American females between the ages of 21 and 60
  Interventions: Other: Survey of exercise practices

INTERVENTIONS:
Other: Survey of exercise practices — detailed questionnaire regarding the subject's race, income level; type(s), frequency, intensity, and amount of exercise; attitudes about exercise; hair style; hair care practices; attitudes about hair; hair and scalp health; and attitudes about exercise with regards to hair

SUMMARY:
The purpose of this research study is to better understand African American women's hair and hair styling practices and how these practices affect attitudes and viewpoints regarding exercise.

ELIGIBILITY:
Inclusion Criteria:

* Female between 21 and 60 years old.
* African, Afro-Caribbean, or African American decent.
* Able and willing to follow study procedures and successfully complete hair and exercise questionnaire/survey.

Exclusion Criteria:

* Unable to read or understand hair and exercise questionnaire/survey.

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: African American females between the ages of 21 and 60.These subjects will be recruited from Wake Forest University Health Sciences Dermatology clinic and our Institutional Review Board (IRB) approved advertising.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2007-09-19 (Actual); Primary Completion 2013-01-30 (Actual); Study Completion 2013-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy McMichael, MD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No